CLINICAL TRIAL: NCT04674670
Title: The Role of Dopamine in Fronto-striatal Activation in Emotional-motivational Pain Processing in Patients With Chronic Pain
Brief Title: Psychobiological Mechanisms Underlying Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: susanne becker (Other)
Collaborators: SNSF (Unknown)
Responsible Party: Sponsor-Investigator, susanne becker, Head of Research Group, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PR00P1_179697/1_3_4
Record Dates: First submitted 2020-12-03; First posted 2020-12-19 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Fibromyalgia; Pain, Chronic; Chronic Pain, Widespread
Keywords: Fibromyalgia; acute pain; chronic pain; Widespread Pain; hedonic shift; Dopamine; Magnetic Resonance Imaging; Functional connectivity; emotional-motivational components of pain; sensory-discriminative components of pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Acute Pain | interventions — Bromocriptine; Amisulpride

STUDY DESIGN:
Intervention Model Description: The drugs that will be used in this study will not be utilised as therapeutic clinical interventions, but as modulators of endogenous process and to assess psychobiological mechanisms in pain processing. Healthy controls will be administered with placebo or a dopamine agonist (bromocriptine) or a dopamine antagonist (amisulpride) on separate days to investigate the role of dopamine and fronto-striatal functional connectivity and BOLD response in relation to emotional-motivational component of pain. Fibromyalgia patients receive only placebo or a dopamine agonist to see the effects of normalization of dopamine on fronto-striatal connectivity and BOLD response, because a lowered dopamine level is assumed to decrease the emotional-motivational component of pain.
Who Masked: Participant, Investigator
Masking Description: Double-blinded randomized placebo-controlled between-within-subject cross-over design with repeated measures; Participants and experimenter will be blinded through out the complete data collection. In addition, participants are not fully instructed about the purpose of the specific tests during the test session, but will be debriefed after final testing session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy controls (Experimental): In this arm, healthy controls will be administered placebo or a dopamine receptor agonist or a dopamine receptor antagonist on separate days to investigate the role of dopamine and fronto-striatal functional connectivity and BOLD response in relation to emotional-motivational pain processing.
  Interventions: Drug: Bromocriptine Mesylate Capsules; Drug: Amisulpride 400 MG; Drug: Placebo
- Fibromyalgia patients (Experimental): In this arm, fibromyalgia patients will receive placebo or a dopamine receptor agonist to investigate the effects of normalizing dopamine transiently on fronto-striatal connectivity and BOLD response in relation to emotional-motivational pain processing.
  Interventions: Drug: Bromocriptine Mesylate Capsules; Drug: Placebo

INTERVENTIONS:
Drug: Bromocriptine Mesylate Capsules — Healthy controls and fibromyalgia patients will be administered a single dose of bromocriptine (1.25mg, p.o.) to investigate the effect of transiently increasing the availability of dopamine on fronto-striatal functional connectivity and BOLD response in relation to emotional-motivational pain processing.
Drug: Amisulpride 400 MG — Healthy controls will be administered a single dose of amisulpride (400mg, p.o.) to investigate the effect of transiently decreasing the availability of dopamine on fronto-striatal functional connectivity and BOLD response in relation to emotional-motivational pain processing.
  Arms: Healthy controls
Drug: Placebo — Healthy controls and fibromyalgia patients will be administered a placebo as for comparison with the effects of bromocriptine (healthy controls and patients) and amisulpride (healthy controls only) on fronto-striatal functional connectivity and BOLD response in relation to emotional-motivational pain processing.
  Other Names: Placebo for substudy 2

SUMMARY:
Pain is a powerful motivator of behavior and it is more than the perception of nociceptive input. It is a complex experience that comprises different components: sensory discriminative, emotional-motivational and cognitive components. In chronic pain, a negative hedonic shift has been proposed that is characterized by disproportionally increased emotional-motivational compared to sensory-discriminative pain components. Such a negative hedonic shift is mirrored in a high comorbidity of chronic pain with affective disorders like depression and anxiety. However, the neurobiological mechanisms underlying such a negative hedonic shift i remain elusive. Animal work suggests an involvement of neuroinflammation, caused by chronic pain, which in turn is related to impaired release of the neurotransmitter dopamine. In line with this observation, impaired dopamine functioning has been described in chronic pain. Importantly, dopamine acts also as a neuromodulator, regulating functional connectivity between brain regions. Therefore, dysfunctional dopamine in chronic pain, possibly caused by neuroinflammation, might lead to altered blood oxygen level dependent (BOLD) response and functional connectivity. Correspondingly, altered functional connectivity in fronto-striatal brain networks has been shown to be predictive of transition from subacute to chronic pain. The aim of this study is to investigate the psychobiological mechanisms underlying the negative hedonic shift in chronic pain with a focus on the role of dopamine in functional connectivity of fronto-striatal brain networks, BOLD response of frontostriatal regions and their relation to heightened emotional-motivational pain processing.

DETAILED DESCRIPTION:
Pain is a powerful motivator of behavior and it is more than the perception of nociceptive input. It is a complex experience that comprises different components: sensory discriminative, emotional-motivational and cognitive components. In chronic pain, a negative hedonic shift has been proposed that is characterized by disproportionally increased emotional-motivational compared to sensory-discriminative pain components. Such a negative hedonic shift is mirrored in a high comorbidity of chronic pain with affective disorders like depression and anxiety. However, the neurobiological mechanisms underlying such a negative hedonic shift remain elusive. Animal work suggests an involvement of neuroinflammation, caused by chronic pain, which in turn is related to impaired release of the neurotransmitter dopamine. In line with this observation, impaired dopamine functioning has been described in chronic pain. Importantly, dopamine acts also as a neuromodulator, regulating functional connectivity between brain regions. Therefore, dysfunctional dopamine in chronic pain, might lead to altered functional connectivity. Correspondingly, altered functional connectivity in fronto-striatal brain networks has been shown to be predictive of transition from subacute to chronic pain. The aim of this study is to investigate the psychobiological mechanisms underlying the negative hedonic shift in chronic pain with a focus on the role of dopamine in functional connectivity of fronto-striatal brain networks, BOLD response of frontostriatal regions and their relation to heightened emotional-motivational pain processing.

A potential benefit of the study will be an increase in our knowledge on mechanisms of the development and maintenance of chronic pain in humans with a focus on emotional-motivational processes, deemed to be of very high relevance in this context. Importantly, by implementing and testing a novel conceptual framework, the results will be relevant not only to pain research but also to a broader neuroscientific community, because the expected results also relate to affective and motivational processes in other diseases (e.g. depression, anxiety, Parkinson's disease). The proposed project offers novel avenues to pain treatment based on pharmacological and psychological mechanisms-based approach instead of being symptoms-oriented as most available pain treatments at the moment.

This study entails more than minimal risks and burdens for participants, because the study incorporates the intake of drugs. However, the study requires only low doses and/or single doses of the drug. In this study, patients with fibromyalgia and healthy participants will receive a single dose of the dopamine agonist bromocriptine (1.25 mg, p.o.) or a placebo in separate testing sessions. Healthy participants will receive in an additional testing session a single dose of the dopamine antagonist amisulpride (400 mg, p.o.). Both drugs have been repeatedly used in research with the same dosages with no or very few side effects. The methods that will be used in the experimental testing sessions are within the range of standard procedures in pain research and experimental psychology and are frequently used in healthy participants and patients. Experimental pain stimulation will be adjusted to individual pain sensitivity, rendering the applied stimulation tolerable. Magnetic resonance imaging will be performed without a contrast medium. Peripheral venous blood sampling will be performed by an expert medical professional. The risk of unauthorized data access or unwanted identification of participants will be minimized by the use of restricted access to data and facilities, lockable cabinets, and password protected computers.

The sample consists of fibromyalgia patients and age- and sex-matched healthy controls. While healthy controls undergo three testing sessions to assess the effects of a dopamine receptor antagonist and agonist in comparison to placebo, fibromyalgia patients perform only two testing sessions assessing only the effects of a dopamine agonist in comparison to a placebo, because for these patients the presence of a hypodopaminergic state is assumed. Thus, each session comprises the intake of a single dose of a drug or placebo and MRI scanning. Healthy controls will take in amisulpride (dopamine receptor antagonist), bromocriptine (dopamine receptor agonist), and placebo and fibromyalgia patients bromocriptine and placebo in a counterbalanced order. At the beginning of the first session, written consent will be obtained from the participants after explaining them the purpose and the course of the experiment. After intake of the capsules containing drug/placebo, there will be a waiting period to reach the peak plasma concentration of the drugs during MRI scanning. During this waiting period, participants will fill out some questionnaires. Before the MRI scanning, in each testing session, pain assessments will be performed, which includes assessment of participants individual heat pain threshold and tolerance. This will be followed by taking a blood sample to determine prolactin levels, pro-inflammatory cytokines and anti-inflammatory cytokines and neurofilaments, after which participants will be positioned inside the MRI scanner. During MRI scanning, participants will perform a behavioral discrimination task and an avoidance task to assess sensory-discriminative and emotional-motivational pain components. After completion of these tasks, resting state fMRI will be performed followed by a structural MRI acquisition for obtaining anatomical images. The duration for each testing session is 3-3.5h.

Sample sizes are based on a priori sample size calculations using G*Power 3.1 with a desired medium effect size f= 0.25, alpha = 0.05, beta= 0.95, repeated measures ANOVA within-between subject designs, and an attrition rate of 10%. Outcome variables will be analyzed in separate mixed model analyses for ANOVA designs with appropriate within- and between-subject factors. Associations of primary endpoints with questionnaire scores (secondary outcomes) will be analyzed using Pearson- or Spearman correlation coefficients, where appropriate. Significance levels will be set to 5%, adjusted with false discovery rate for multiple testing. Effect sizes will be calculated in terms of generalized eta-squared (ηG2) and Cohen's d. Images from fMRI analysis of each participant will undergo standard preprocessing (including high-pass filtering, motion correction, spatial smoothing) and will be entered into a voxel-wise analysis using a general linear model to estimate the effects of pharmacological interventions on pain-related brain activity related to emotional-motivational and sensory-discriminative pain responses. For all brain analyses, a voxel-threshold of p<0.01 and a cluster threshold for spatial extent of p<0.05 will be employed.

Within this study, pharmacological interventions, psychophysical methods, and magnetic resonance imaging will be utilized to investigate the neurobiological mechanisms involved in a negative hedonic shift in chronic pain. Pharmacological interventions (amisulpride and bromocriptine) will only cause a transient manipulation of dopaminergic system in both healthy controls and fibromyalgia patients. The pharmacological interventions proposed in the current study does not have a clinical intervention value, instead they are only used for the purpose of investigating psychobiological mechanisms underlying chronic pain. Psychophysical methods will allow the investigators to dissociate the emotional-motivational component of pain from its sensory discriminant component. Magnetic resonance imaging will allow the investigators to investigate brain responses and neuroinflammation in relation to chronic pain. Based on these methods, the investigators will get insights on the role of dopamine and fronto-striatal BOLD response and connectivity in regulating the emotional component of pain in chronic pain. The usage of the pharmacological interventions in this study hold more than minimal risks for the participants, but according to previous research studies, in which the same dosage of these pharmacologic drugs were used, only minimal side-effects have been observed (see above "Risk/Benefit Assessment"). Psychophysical methods and pharmacological interventions based on experimental psychology and pain research will be used in this study. These methods have been shown to be successful in investigating the different aspects of pain perception and modulation of pain perception. The methods used are in the standard range of methods from human pain research and experimental psychology. The expected results will form the basis for the development of novel mechanism-based pain therapies.

ELIGIBILITY:
For fibromyalgia patients:

Inclusion criteria:

* Age between 18 to 70 years
* Chronic widespread pain
* Symptoms such as fatigue, cognitive dysfunction, and/or depressive symptoms
* Sufficient knowledge of German or English to follow instructions
* Ability to give written informed consent

Exclusion criteria:

* Psychiatric or neurological disorders, except depression and anxiety
* Substance abuse or consumption of alcohol, illegal drugs, analgesics apart from prescribed routine medication within the last 24 h before testing session
* Pacemaker or metal parts in the body or any contradictions to MRI
* Pregnancy and breast-feeding
* Medical history indicating any risk/allergies using the amisulpride or bromocriptine or both or other ergotamine. Long QT syndrome, cardiac arrhythmia, intake of drugs causing QT prolongation in the electrocardiogram.
* Liver or/and kidney problems
* High blood pressure or cardiovascular or heart disease
* Stomach ulcers or bleeding
* Fibrosis
* Diabetes
* Cancer patients
* Intake of drugs lowering potassium levels in the blood
* Blood pressure problems during pregnancy in the past
* History of breast cancer in the family first-order relatives
* Cerebrovascular events in anamnesis
* Simultaneous intake of potent or moderate Cytochrome P450 inhibitors

For Healthy participants:

Inclusion criteria:

* Age-matched healthy participants
* Good overall health status
* Sufficient knowledge of German or English to follow instructions
* Ability to give written informed consent

Exclusion criteria:

* Pain longer than 3 consecutive days and on more than 30 days within the last 12 months
* Major psychiatric or neurological disorders
* Pregnancy and breast-feeding
* Substance abuse or consumption of alcohol, illegal drugs, and analgesic drugs within 24 h before testing session
* Pacemaker or metal parts in the body or any contradiction to MRI
* Medical history indicating any risk/allergies using the amisulpride or bromocriptine or both or other ergotamine.
* Liver or/and kidney problems
* High blood pressure or cardiovascular or heart disease
* Stomach ulcers or bleeding
* Fibrosis
* Diabetes
* Low potassium levels in the blood
* Blood pressure problems during pregnancy in the past
* History of breast cancer in first-order relatives
* Cerebrovascular events in anamnesis
* Simultaneous intake of potent or moderate Cytochrome P450 inhibitors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level dependent (BOLD) responses | approx. 90 minutes
  blood oxygen level dependent (BOLD) signal variance (%) from the baseline
Sensory pain responses | approx. 20 minutes
  correct responses in the task assessing sensory-discriminative pain responses
Emotional pain responses | approx. 20 minutes
  correct responses in task assessing emotional-motivational pain responses

SECONDARY OUTCOMES:
reaction time (RT) | approx. 15 minutes
  reaction times during behavioral tasks
pain threshold | 5 minutes
  Individual pain threshold assessed with experimental heat pain (°C). Participants press the space bar when the temperature start to be painful.
pain tolerance | 5 minutes
  Individual pain tolerance assessed with experimental heat pain. (°C). Participants press the space bar when they cannot tolerate a higher temperature.
perceived pain intensity | approx. 33 minutes
  Individual perceived pain intensity assessed with experimental heat pain. Participants rate the stimuli by moving a cursor with the arrows keys on a scale from 0 (no sensation) to 200 (highest temperature tolerable). The middle of the scale has a mark at 100 (pain threshold).
perceived pain unpleasantness | approx. 33 minutes
  Individual perceived pain unpleasantness assessed with experimental heat pain. Participants rate the stimuli by moving a cursor with the arrows keys on a scale from -100 (extremely unpleasant) to +100 (extremely pleasant). The middle of the scale has a mark at 0 (neutral).
Pain Catastrophizing Scale (PCS) | during the procedure, at day 1
  The PCS was developed in 1995 at the University Centre for Research on Pain and Disability in order to facilitate research on the mechanisms by which catastrophizing impacts on pain experience. Catastrophizing is currently defined as: an exaggerated negative mental set brought to bear during actual or anticipated painful experience.
Beck Depression Inventory (BDI) | during the procedure, at day 1
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression (Beck, et al., 1961). The BDI has been developed in different forms, including several computerized forms, a card form (May, Urquhart, Tarran, 1969, cited in Groth-Marnat, 1990), the 13-item short form and the more recent BDI-II by Beck, Steer & Brown, 1996. (See Steer, Rissmiller & Beck , 2000 for information on the clinical utility of the BDI-II.) The BDI takes approximately 10 minutes to complete, although clients require a fifth - sixth grade reading level to adequately understand the questions (Groth-Marnat, 1990)
Chronic Pain Acceptance Questionnaire - Revised (CPAQ-R) | during the procedure, at day 1
  The 20-item CPAQ-revised has been designed to measure acceptance of pain. The acceptance of chronic pain is thought to reduce unsuccessful attempts to avoid or control pain and thus focus on engaging in valued activities and pursuing meaningful goals.
The Gratitude Questionnaire-Six Item Form (GQ-6) | during the procedure, at day 1
  The Gratitude Questionnaire-Six-Item Form (GQ-6) is a six-item self-report questionnaire designed to assess individual differences in the proneness to experience gratitude in daily life.
Life Orientation Test - Revised (LOT-R) | during the procedure, at day 1
  A 10-item measure of optimism versus pessimism.
State-Trait Anxiety Inventory (STAI form Y-1) | The questionnaire will be filled thrice at three different timepoints in each testing session
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress (e.g., Greene et al., 2017, Ugalde et al., 2014).
Self-Compassion Scale, Short Form (SCS-SF) | during the procedure, at day 1
  Self-compassion entails being kind and understanding toward oneself in instances of pain or failure rather than being harshly self-critical; perceiving one's experiences as part of the larger human experience rather than seeing them as isolating; and holding painful thoughts and feelings in mindful awareness rather than over-identifying with them. Evidence for the validity and reliability of the scale is presented in a series of studies. Results indicate that self-compassion is significantly correlated with positive mental health outcomes such as less depression and anxiety and greater life satisfaction. Evidence is also provided for the discriminant validity of the scale, including with regard to self-esteem measures.
The Resilience Scale (RS-25) | during the procedure, at day 1
  The Resilience Scale (RS25) is an instrument developed by Wagnild and Young (1993) to assess resilience levels in adults. There's seven numbers per items on the scale, ranging from "1" (Strongly Disagree) on the left to "7" (Strongly Agree) on the right. A higher score means a better resilience.
Snaith Hamilton Pleasure Scale (SHAPS) | during the procedure, at day 1
  The SHAPS is a 14-item scale that measures anhedonia, the inability to experience pleasure. The items cover the domains of: social interaction, food and drink, sensory experience, and interest/pastimes. Participants tick one of the boxes to indicate how much they agree or disagree with each statement from 1 (strongly disagree) to 4 (strongly agree). Higher score means a better ability to experience pleasure.
Structured Clinical Interview for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) (SCID-5) | during the procedure, at day 1
  The Structured Clinical Interview for DSM-5 (SCID-5) is a semistructured interview guide for making the major DSM-5 diagnoses. It is administered by a clinician or trained mental health professional who is familiar with the DSM-5 classification and diagnostic criteria. The interview subjects may be either psychiatric or general medical patients-or individuals who do not identify themselves as patients, such as participants in a community survey of mental illness or family members of psychiatric patients.
Fear of Avoidance Beliefs (FABQ) | during the procedure, at day 1
  FABQ focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability
Fear of Pain Questionnaire (FPQ-III) | during the procedure, at day 1
  FPQ-III is one questionnaire which is a widely used to assess the fear of pain (FOP) in clinical and non clinical samples. It is one self-report instrument that was developed specifically to assess fear of different stimuli usually causing pain.
The Need Inventory of Sensation Seeking (NISS) | during the procedure, at day 1
  The Need Inventory of Sensation Seeking (NISS) by Roth and Hammelstein (2012) conceptualizes sensation seeking as a motivational trait, a need for stimulation that can provoke different behaviors.
Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking, Positive Urgency, Impulsive Behavior Scale (UPPS-P, Short version) | during the procedure, at day 1
  The UPPS-P model of impulsivity proposes that impulsivity as a multi-faceted and multi-dimensional construct, comprising five impulsive personality traits.
Big Five Personality Traits Questionnaire | during the procedure, at day 1
  It measures the big five dimensions of personality
West Haven-Yale multidimensional pain inventory - Part A | during the procedure at day 1
  Components of chronic pain experience are assessed using this questionnaire
Positive and Negative Affect Schedule (PANAS) | during the procedure, at day 1, day 2 and day 3
  Mood will be assessed using PANAS
Emotion Regulation Questionnaire | during the procedure, at day 1
  It is a 10-item scale which measures the tendency of the participant to regulate their emotions.
Prolactin and Estradiol | during the procedure, at day 1, day 2 and day 3
  Concentration of prolactin and estradiol will be identified in collected blood samples
Pro-inflammatory and anti-inflammatory cytokines | during the procedure, at day 1
  Concentration of cytokines will be identified in collected blood samples using U-PLEX MSD multiplexing panel
Neurofilament Analysis | during the procedure, at day 1
  Concentration of Neurofilament will be than determined with a new-generation automatised immunoassay method, the simple plex ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Becker, PD Dr., Principal Investigator — Balgrist Universitätsklinik
Locations (1):
- Balgrist Campus, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No